CLINICAL TRIAL: NCT03252366
Title: MAXILLARY SINUS ELEVATION USING GELFOAM (ABSORBABLE GELATIN) VERSUS XENOGRAFT (TUTOGEN) and SIMULTANEOUS IMPLANT PLACEMENT:Randomized Clinical Trial
Brief Title: Maxillary Sinus Elevation and Simultaneous Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, fatma fawzy kandel, Master degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MI.cairouniversity
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Maxillary Sinus
Keywords: MAXILLARY SINUS ELEVATION ,Simultaneous implant placement
MeSH Terms: interventions — Gelatin Sponge, Absorbable; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GELFOAM (ABSORBABLE GELATIN) (Active Comparator): Sterile Sponge is a medical device intended for application to bleeding surfaces as a hemostatic. It is a water-insoluble, off-white, nonelastic.
  it act as a space maintainer and alternative to bone filler for new bone formation in the maxillary sinus. It may be cut without fraying and is able to absorb and hold within its interstices, many times its weight of blood and other fluids its effect appears to be more physical than the result of altering the blood clotting mechanism. When placed in soft tissues, GELFOAM is usually absorbed completely within four to six weeks, without inducing excessive scar tissue
  Interventions: Device: GELFOAM
- XENOGRAFT (TUTOGEN) (Active Comparator): xenografts as a sinus bone replacement graft ,The osteoconductive properties of xenografts in human sinus grafting have been well documented. They are due to both their chemical composition and their macro and micro morphology.The efficacy of xenografts as a sinus bone replacement graft may be due to combination of factors. Foremost would be the osteoconductive capacity of xenografts. In addition, they supply minerals that are necessary for bone formation, their density provides stability to the graft and the implants placed in them, and this density persists long term due to the fact that these grafts do not completely resorb.
  Interventions: Device: xenograft

INTERVENTIONS:
Device: GELFOAM — * Three line mucoperiosteal pyramidal flap will be reflected in the posterior maxillary edentulous area to expose the lateral wall of the maxilla.
  * A diamond bur will be used to make a rectangular osteotomy.
  * The membrane will be carefully elevated from the lateral wall and floor of maxillary sinus with simultaneous implant placement.
  * Implant stability will be measured by osteal device
  * implant will be inserted with gelfoam (absorbable gelatin) for augmentation• The flap will then be copiously irrigated with saline in preparation for closure.
  * The flap will then be closed using interrupted 4/0 resorbable sutures.
  Other Names: (ABSORBABLE GELATIN)
  Arms: GELFOAM (ABSORBABLE GELATIN)
Device: xenograft — * Three line mucoperiosteal pyramidal flap will be reflected in the posterior maxillary edentulous area to expose the lateral wall of the maxilla.
  * A diamond bur will be used to make a rectangular osteotomy.
  * The membrane will be carefully elevated from the lateral wall and floor of maxillary sinus with simultaneous implant placement.
  * Implant stability will be measured by osteal device
  * implants will be inserted with xenograft for augmentation.• The flap will then be copiously irrigated with saline in preparation for closure.
  * The flap will then be closed using interrupted 4/0 resorbable sutures.
  Other Names: TUTOGEN
  Arms: XENOGRAFT (TUTOGEN)

SUMMARY:
using gel foam [ absorbable gelatin ] in maxillary sinus elevation which act as a space maintainer and alternative to bone filler for new bone formation in the maxillary sinus and its advantages for patients undergoing maxillary sinus elevation with simultaneous implant placement as regards the implant stability and amount of bone height gain compared to conventional maxillary sinus elevation by xenograft.

DETAILED DESCRIPTION:
One of the main problem for posterior maxilla it becomes atrophic after extraction of the teeth and this followed by Pneumatization of the maxillary sinus, the atrophy of the alveolar process is a common reason for the limited availability of alveolar bone for implant placement in the posterior maxilla.

Numerous techniques designed to increase bone volume in the maxillary sinus region have been proposed. They were mostly based on the insertion of various materials into a void created between the sinus (Schneiderian) membrane and the bony walls of the maxillary sinus. (Sohn et al 2008) reported simultaneous placement of implants, and insertion of gelatin sponges demonstrate new bone formation through clinical and radiographic evaluations. New bone formation was verified by stabilization of the elevated sinus membrane from the tenting effect of placement of dental implants and absorbable gelatin sponge without any bone graft material. This study shows that there is great potential for new bone formation in the maxillary sinus without the use of additional bone grafts. Systemic review showed that the survival rate for implants utilizing xenografts was statistically the same as for implants placed in particulate autogenous bone grafts .

ELIGIBILITY:
Inclusion Criteria:• Patients with atrophic maxilla and pneumatization of the maxillary sinus with residual bone height from 3 to 5mm .

* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:• Sinus pathology.

* Heavy smokers more than 20 cigarettes per day .
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems.
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Amount of bone gained: | 6 month
  using linear measurements from Cone beam computed tomography

IPD SHARING:
Plan to Share IPD: Undecided